CLINICAL TRIAL: NCT07036289
Title: Effects Of PeriodontitisTtreatment On The Worsening Of Heart Failure: A Randomized Clinical Trial
Brief Title: Periodontitis Treatment and Heart Failure
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Taubate (Other)
Collaborators: Federal University of Minas Gerais (Other); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Jose Roberto Cortelli, dentist, specialist, master and doctorate, University of Taubate
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAAE 76621623.3.00000.5501; 2023/07458-4 (Other Grant/Funding Number: FAPESP); 306161/2023 (Other Grant/Funding Number: CNPQ)
Record Dates: First submitted 2025-06-14; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Heart Failure; Periodontitis
Keywords: scaling and root planing; heart failure; periodontitis; NT-proBNP; saliva; blood; Porphyromonas Gingivalis
MeSH Terms: conditions — Heart Failure; Periodontitis

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: statistics and laboratorial exams personnel
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- periodontitis heart failure mechanical treatment (Experimental): scaling and root planing plus oral hygiene instructions
  Interventions: Procedure: Mechanical Treatment
- periodontitis mechanical treatment (Active Comparator): scaling and root planing plus oral hygiene instructions
  Interventions: Procedure: Mechanical Treatment
- periodontitis heart failure control (No Intervention): oral hygiene instructions

INTERVENTIONS:
Procedure: Mechanical Treatment — manual quadrant scaling and root planing followed by dental prophylaxis within 4 weekly sections and oral hygiene instructions
  Arms: periodontitis heart failure mechanical treatment; periodontitis mechanical treatment

SUMMARY:
Heart failure (HF) is a rapidly growing public health issue affecting more than 40 million individuals globally; while gum disease with bone loss affects 50% of people in general. The objective of this study is to evaluate the effect of dental treatment on blood levels of a HF parameter at 3 and at 6 months. In addition to verify the relation between blood and salivary exam results and severity of HF. Imune response against one important oral bacterial will be also monitored at 3 and 6 months. Approximately 80 adult individuals will be included and divided into 3 groups. The first two groups will receive dental scaling and root planing (periodontitis individuals with heart failure [n = 25]; periodontitis individuals without heart failure [n = 25]). The third group named negative control will receive dental treatment only after 6 months of dental follow-up (periodontitis individuals with heart failure [n = 25]). HF treatment by oral medication will be continuous. Blood, salivary, microbiological and immune examinations will be performed in addition to the periodontal treatment of scaling and root planning. Clinical data will be obtained both for initial diagnosis and disease staging and for longitudinal follow-up.

DETAILED DESCRIPTION:
Heart failure (HF) is a rapidly growing public health issue with an estimated prevalence of > 40 million individuals globally; while periodontitis affects 50% of people in general, and its most severe form affects approximately 11% of the population. The primary objective of this study is to evaluate the effect of periodontal therapy on blood levels of NT-proBNP (N-terminal pro-B-type natriuretic peptide) at 3 and at 6 months. Secondary aims are the relation between biomarker blood levels and a) functional classes and b) its salivary levels. Antibodies against P. gingivalis besides species' levels will be also determined initially and at 3 and 6 months. As 66 participants must complete the study, 75 to 85 individuals over 35 years of age will be included and randomly assigned to dental scaling and root planing (periodontitis individuals with heart failure [n = 25]; periodontitis individuals without heart failure [n = 25]) or negative control (periodontitis individuals with heart failure [n = 25]). Blood, salivary, microbiological and immune examinations will be performed in addition to the periodontal treatment of scaling and root planning. Clinical data will be obtained both for initial diagnosis and disease staging and for longitudinal follow-up. NT-proBNP and antibodies against P. gingivalis will be evaluated by enzyme immunoassay using commercially available kits while P. gingivalis levels will be determined by quantitative polymerase chain reaction (qPCR).

ELIGIBILITY:
Inclusion Criteria:

* minimum of 35 years of age;
* possibility and availability for medical and dental examinations;
* specifically for HF groups: HF having as primary causes ischemic problems, myocardial infarction, hypertension and valvulopathies will be selected
* HF with intermediate or reduced ejection fraction under one of the three following pharmacological therapeutic regimens: a) Angiotensin Converting Enzyme Inhibitors, as the first option, or b) Angiotensin II Receptor Blockers and b) Angiotensin II Receptor Blockers and c) Angiotensin/neprilysin receptor inhibitors.

Exclusion Criteria:

* pregnant or lactating women;
* individuals with stage D of HF using vasoactive drugs or circulatory devices;
* HF individuals with preserved ejection fraction;
* participants who do not meet the criteria for periodontal disease;
* participants who are unable to comply with the study protocol;
* diabetes, obesity, chronic kidney disease and other non-ischemic causes of HF;
* familial and congenital heart alterations and myocarditis
* rheumatological and autoimmune diseases;
* drugs and cardiotoxic substances such as cocaine and oncological chemotherapy;
* Specifically for the negative control group a progression of periodontitis revealed by 0.3mm additional clinical attachment loss within 6 months of follow-up.

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2025-06-10 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
NT-proBNP in blood samples | baseline versus 6 months
  Changes in NT-proBNP (N-terminal pro-B-type natriuretic peptide) levels in blood samples. Higher levels indicate worse heart failure status.

SECONDARY OUTCOMES:
Salivary NT-proBNP | baseline, 3 and 6 months
  Comparative NT-proBNP levels between blood and saliva samples at each time-point
clinical pocket depth response | baseline, 3 and 6 months
  Changes in periodontal pocket depth (mm). Higher values indicate deeper periodontal pockets.
clinical attachment level response | baseline, 3 and 6 months
  Changes in periodontal clinical attachment level (mm). Higher values indicate worse periodontal breakdown.
clinical bleeding response | baseline, 3 and 6 months
  Changes in bleeding on probing (0 indicates absence and 1 presence of bleeding onto gentle periodontal probing).
P. gingivalis bacterium salivary levels | baseline and 3 months
  P. gingivitis bacterium levels in saliva samples
P. gingivalis antibody salivary levels | baseline and 3 months
  Antibodies against P. gingivitis in saliva samples

CONTACTS AND LOCATIONS:
Overall Officials: Jose R Cortelli, Doctorate, Principal Investigator — University of Taubate
Locations (1):
- University of Taubate Dental School, Taubaté, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
Data will be analyzed by blind statistics and laboratorial staff and there is no need for sharing IPD.